CLINICAL TRIAL: NCT00469352
Title: The Effect of Genotype and Environmental Risk Factors on Treatment Response to Intravitreal Lucentis (Ranibizumab) for Neovascular AMD
Brief Title: A Study of Genetic and Environmental Factors and Their Effect on Response to Treatment With Lucentis (Ranibizumab) for Wet AMD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Peter Francis, MD, PhD, Oregon Health & Science University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00003335
Record Dates: First submitted 2007-05-02; First posted 2007-05-04 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Macular Degeneration
Keywords: Pharmacogenetics; Genetics; Treatment response; AMD; Wet AMD; Age-related macular degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ranibizumab — Ranibizumab as needed

SUMMARY:
The purpose of this study is to understand whether genes or certain factors in the environment determine how eyes will respond to Lucentis (ranibizumab) treatment. For example, whether having variants within specific genes means that a patient is likely to get better vision from treatment than another patient with different genes.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is the leading cause of blindness in the developed world. The advanced stages of the disease are characterized by the development of geographic atrophy or choroidal neovascularization, both of which result in significant loss of vision. Development of intravitreal anti-VEGF agents such as ranibizumab has significantly improved outcomes for the neovascular for of the disease. However, it is not possible to predict which individuals will respond to the treatment.

The objective of this study is to establish the association between genetic factors and treatment response to intravitreal Lucentis. This will be accomplished by SNP-genotyping participants for AMD-susceptibility and candidate angiogenesis-pathway genes, collecting environmental risk factor variables and evaluating clinical outcomes. The aim of this pharmacogenetics study will be to identify patients at the outset of their treatment that require more intensive therapy.

ELIGIBILITY:
Inclusion Criteria:

* All AMD-related CNV lesion types will be included.
* Age >50 years
* The study eye must never have received treatment for neovascular AMD
* Visual acuity in treatment eye must be between 20/30 and 20/320 (ETDRS).

Exclusion Criteria:

* Age <50 years;
* Previous therapy in either eye for AMD or other retinal disease which may be used in the treatment of AMD;
* Choroidal neovascularization not from AMD;
* Concomitant non-AMD related maculopathy in study eye;
* Active treatment for neovascular AMD in fellow eye;
* Acuity loss or central field loss from non-AMD cause;
* Pigment epithelial detachment without evidence of CNV;
* Individuals in whom Lucentis is contraindicated;
* Participation in another clinical trial in last three months
* Pregnancy (positive pregnancy test) or lactation
* Premenopausal women not using adequate contraception
* Prior enrollment in the study
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2007-05; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is clinical treatment response to intravitreal Lucentis, defined as: 'Clinical stabilization' : stabilization of visual acuity. 'Clinical improvement'; 'Clinical progression' | 12 months

SECONDARY OUTCOMES:
Establish the association between environmental risk factors and treatment response to intravitreal Lucentis when controlling for genotype | 12 months
Association between central macular thickness as measured by ocular coherence tomography (OCT) in response to Lucentis treatment and genotype/environmental risk exposure. | 12 months
Median number of intravitreal ranibizumab (Lucentis) injections required per patient | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Francis, MD PhD, Principal Investigator — Casey Eye Institute, Oregon Health and Science University
Locations (1):
- Casey Eye Institute, Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- [Derived] Francis PJ. The influence of genetics on response to treatment with ranibizumab (Lucentis) for age-related macular degeneration: the Lucentis Genotype Study (an American Ophthalmological Society thesis). Trans Am Ophthalmol Soc. 2011 Dec;109:115-56. PMID 22253485